CLINICAL TRIAL: NCT01150071
Title: Growth, Health and Development in Children Born Extremely Preterm
Acronym: PEP11
Status: Completed | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Trond Markestad, Professor, University of Bergen
Other Study IDs: 2009/2271-1
Record Dates: First submitted 2010-06-23; First posted 2010-06-24 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Infant, Extremely Low Birth Weight; Lung Diseases, Obstructive; Disorder of Bone Density and Structure, Unspecified; Cognition Disorders; Neurobehavioral Manifestations
Keywords: extremely premature infant; follow-up; behavior; growth; mental health; lung function; spirometry; muscle mass; bone density; magnetic Resonance imaging
MeSH Terms: conditions — Lung Diseases, Obstructive; Cognition Disorders; Neurobehavioral Manifestations; Behavior; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — On a subpopulation blood for inflammatory parameters will be collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children born extremely preterm: national cohort of children born before 28 weeks' gestational age or with a birthweight less than 1000 g. 365 eligible survivors

SUMMARY:
Background: In a national Norwegian cohort of children born before 28 weeks gestation or with a birth weight less than 1000 g born in 1999 and 2000, 372 survived. Compared with earlier studies survival increased for the most immature infants, but at the cost of more early complications and a high rate of impairments, while the less immature children had fewer early complications and less impairments detectable within 5 years. These changes show the importance of monitoring outcome as treatment modalities change. Large brain haemorrhages were highly predictive of severe disabilities, but we have not found good predictive factors for milder impairments such as cognitive, behavioural and motor difficulties. However, at 5 years later function may be difficult to predict, and the children's potentials are better understood after completing several years in school. Objectives: The children will be re-examined at age 11 in order to assess their physical and mental health, and cognitive, motor and social function, and to determine if early life events and development at 2 and 5 years are predictive of long term health and functioning. MRI-studies, including functional MRI will be performed to examine if different outcomes related to brain function can be explained by differences in brain development. Methods: For all, data will be collected from the compulsory national test in 5th grade and questionnaires to the child, parents and teacher. For children in Western Norway (n=87) extensive examinations of lung and brain function, including clinical diagnostic tests and MRI, will be added. For all aspects of the study the investigators have appropriate current and historic reference populations for comparison. Implications: Knowledge on causes and of early predictions of outcome is needed to give appropriate advice to families, professionals and society, and to develop preventive programs.

DETAILED DESCRIPTION:
Questionnaires to parents: On general and neurosensory developmental Health (spesific questionnaire for the study) and pulmonary health (ISAAC-questionnaire). Mental Health and social functioning: Strengths and Difficulties (SDQ) questionnaire (also completed by Teachers), ASSQ and BRIEF.

Addtions for children born in the Western Norway Regional Health Authority:

All the children (n=52) and matched Controls born at term have measurements of height, weight and blood pressures, pulminary function tests, MRI and functional MRI of the brain, Assessment of bone mineralization and distribution of fat and muscle (DXA). Blood is collected in a biobank for assessment of inflammatory variables.

ELIGIBILITY:
Inclusion Criteria:

* Born in 1999 and 2000 with gestational age < 28 weeks or birth weight < 1000 g
* still living when 11 years old

Exclusion Criteria:

* None

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All extremely preterm infants (gestational age < 28 weeks or birth weight < 1000 g born in Norway in 1999 and 2000 and still living at age 11 years. Postal survey on outcome. In addition a subgroup (80 out of 365)living in Western Norway will be examined with respect to general health, lung function, mental development, quality of life and cerebral imaging (fMRI)
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
growth | Eleven years old (years 2010, 2011)
  Heigh and weight. In a subpopulation of 80 children: Also skin fold thicknesses and waist circumference
Mental health | Eleven years old (years 2010, 2011)
  Questionnaires completed by parents (Strengths and Difficulties questionnaire, Parenting Stress Index,ASSQ)
Cognitive function | Eleven years old (years 2010, 2011)
  Grades in 5th grade in school
Pulmonary function | Eleven years of age (years 2010,2011)
  Spirometry on a subgroup of 80 and 80 controls
Cerebral function | Eleven years of age (years 2010,2011)
  fMRI on a subgroup of 40 and 40 controls
Bone density | Eleven years of age (years 2010,2011)
  DXA measurements on a subgroup of 80 and 80 controls

CONTACTS AND LOCATIONS:
Overall Officials: Trond Markestad, MD, PhD, Principal Investigator — University of Bergen, Faculty of Medicine
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Stavanger University Hospital, Stavanger